CLINICAL TRIAL: NCT06500026
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With Topotecan in Patients With Recurrent Small Cell Lung Cancer After Failure of Anti-PD-1/PD-L1 Monoclonal Antibodies and Platinum-based Chemotherapy
Brief Title: A Study Comparing BL-B01D1 With Topotecan in Patients With Recurrent Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-304
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Topotecan (Experimental): Participants receive Topotecan as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Topotecan — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Topotecan

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with recurrent small cell lung cancer after failure of anti-PD-1/PD-L1 Monoclonal Antibodies and platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Age ≥18 years old;
3. Expected survival time ≥3 months;
4. Patients with recurrent small-cell lung cancer after failure of anti-PD-1/PD-L1 monoclonal antibodies and platinum-based chemotherapy;
5. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
6. Must have at least one measurable lesion according to RECIST v1.1 definition;
7. ECOG 0 or 1;
8. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
10. The organ function level must meet the requirements on the premise that blood transfusion is not allowed within 14 days before the screening period, and no cell growth factor drugs are allowed;
11. A serum pregnancy test must be performed within 7 days before the start of treatment for premenopausal fertile women, and the result must be negative and must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. The patient has histological or cytologic evidence of non-small cell lung cancer or mixed components of small cell lung cancer/non-small cell lung cancer;
2. Prior to randomization, chemotherapy, targeted therapy, or biological therapy were used within 4 weeks or 5 half-lives, small molecule targeted therapy was used within 5 days, or palliative radiotherapy was used within 2 weeks;
3. Patients with recurrent small cell lung cancer who are eligible for curative local therapy;
4. Received chemotherapy with TOP I inhibitor;
5. Received anti-EGFR and/or HER3 antibody /ADC drugs;
6. History of severe heart disease or cerebrovascular disease;
7. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
8. Complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
9. Diagnosis of active malignancy within 3 years before randomization;
10. Hypertension poorly controlled by two antihypertensive drugs;
11. Patients with poor glycemic control;
12. A history of ILD requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis;
13. Complicated pulmonary diseases leading to clinically severe respiratory function impairment;
14. Patients with active central nervous system metastases;
15. Severe infection within 4 weeks before randomization; There was evidence of pulmonary infection or active pulmonary inflammation requiring clinical intervention within 2 weeks before randomization;
16. Patients with massive or symptomatic effusions or poorly controlled effusions;
17. Imaging examination showed that the tumor had invaded or enveloped the large blood vessels in the abdomen, chest, neck, and pharynx;
18. Severe unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
19. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
20. Patients with inflammatory bowel disease, extensive bowel resection history, immune enteritis history, intestinal obstruction, chronic diarrhea or Gilbert's syndrome;
21. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of BL-B01D1;
22. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
23. A history of severe neurological or mental illness;
24. Subjects who were scheduled to receive live vaccine or received live vaccine within 28 days before study randomization;
25. Other circumstances that were assessed by the investigator as inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China